CLINICAL TRIAL: NCT05757011
Title: the Effect of Pre-sacral Nerve Block on Post-operative Pain Following Laparoscopic Hysterectomy: a Triple Blind Placebo Controlled RCT
Brief Title: the Effect of Pre-sacral Nerve Block on Post-operative Pain Following Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Mohamed Mostafa, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MD 247/2020
Record Dates: First submitted 2023-02-20; First posted 2023-03-07 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Gynecology

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Before the removal of uterus and the closure of vaginal cuff, insertion of 6inch 22G needle 2 to 3 cm below the umbilicus, 30 ml normal saline (sodium chloride solution 0.9%, FIPCO, Egypt)will be administered , then the uterus will be removed, and the operation will be terminated
  Interventions: Procedure: pre-sacral nerve block (bupivacaine injection into both uterosacral ligaments at the end of laparoscopic hysterectomy.
- pre-sacral nerve block (Experimental): Uterosacral nerve block will be performed before the removal of uterus and the closure of vaginal cuff, and before the removal of trocars from abdominal cavity, insertion of 6-inch 22G needle 2 to 3 cm below the umbilicus, injection of the SHP area which situated anterior to L5-S1 vertebral bodies, Caudal to the bifurcation of the abdominal aorta with 30 ml 0.25% bupivacaine (Marcaine®0.25% , Astra Zeneca, Egypt) will be administered. Following the injection of local anesthetic, patient will be placed from Trendelenburg position to horizontal position. The we will remove the uterus and trocars , and the operation will be terminated.
  Data will be recorded in a case report form (CRF) and statistical analysis will be done.
  Interventions: Procedure: pre-sacral nerve block (bupivacaine injection into both uterosacral ligaments at the end of laparoscopic hysterectomy.

INTERVENTIONS:
Procedure: pre-sacral nerve block (bupivacaine injection into both uterosacral ligaments at the end of laparoscopic hysterectomy. — pre-sacral nerve block (bupivacaine injection into both uterosacral ligaments at the end of laparoscopic hysterectomy.

SUMMARY:
40 patients who are consenting to be recruited in the study and are fulfilling the eligibility criteria will be subjected to:

Group A Before the removal of uterus and the closure of vaginal cuff, insertion of 6inch 22G needle 2 to 3 cm below the umbilicus, 30 ml normal saline (sodium chloride solution 0.9%, FIPCO, Egypt)will be administered.

While patients randomized to group B will undergo TLH with pre-sacral nerve block.

DETAILED DESCRIPTION:
40 patients who are consenting to be recruited in the study and are fulfilling the eligibility criteria will be subjected to: Group A Before the removal of uterus and the closure of vaginal cuff, insertion of 6inch 22G needle 2 to 3 cm below the umbilicus, 30 ml normal saline (sodium chloride solution 0.9%, FIPCO, Egypt)will be administered , then the uterus will be removed, and the operation will be terminated

While patients randomized to group B will undergo TLH with pre-sacral nerve block as follows:

Uterosacral nerve block will be performed before the removal of uterus and the closure of vaginal cuff, and before the removal of trocars from abdominal cavity, insertion of 6-inch 22G needle 2 to 3 cm below the umbilicus, injection of the SHP area which situated anterior to L5-S1 vertebral bodies, Caudal to the bifurcation of the abdominal aorta with 30 ml 0.25% bupivacaine (Marcaine®0.25% , Astra Zeneca, Egypt) will be administered. Following the injection of local anesthetic, patient will be placed from Trendelenburg position to horizontal position. The we will remove the uterus and trocars , and the operation will be terminated.

Data will be recorded in a case report form (CRF) and statistical analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing elective total laparoscopic hysterectomy Body mass index less than 29 Kg/m2

Exclusion Criteria:

* Previous presacral neurectomy
* Concurrent surgical procedure other than salpingectomy and/or oophorectomy
* Chronic narcotic consumption Inability to provide consent
* Patients with contraindication to laparoscopic surgery (e.g. severe cardiopulmonary dysfunction).
* Bleeding tendency (e.g. patient on anticoagulants, platelets disorders)
* Intra-abdominal adhesions (due to previous abdominal surgery e.g. myomectomy)

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2023-07-10 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
● Post-operative pain 1 hour after the procedure will be assessed by visual analogue scale (VAS). (range will be from zero (no pain) to 10 | 1hour
  ● Post-operative pain 1 hour after the procedure will be assessed by visual analogue scale (VAS). (range will be from zero (no pain) to 10

CONTACTS AND LOCATIONS:
Overall Officials: Gasser Elbishry, Professor, Study Chair — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No